CLINICAL TRIAL: NCT04545216
Title: Assessment of the Impact of an Ultratrail on the Knee Cartilage by Using T2 MRI: a Pilot Study
Brief Title: Impact of Long Distance Mountain Race on Knee Cartilage.
Acronym: UT4M2020
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: UT4M 2020 - 38RC20.008
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Sports Medicine
Keywords: long-distance running; knee cartilage; magnetic resonance imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- UT4M 40: athletes participating to the 40 km mountain race.
  Interventions: Other: Long-distance mountain running
- UT4M 160: athletes participating to the 160 km mountain race.
  Interventions: Other: Long-distance mountain running
- UTV 55: athletes participating to the 55 km mountain race.
  Interventions: Other: Long-distance mountain running

INTERVENTIONS:
Other: Long-distance mountain running — Impact of a mountain race on the knee cartilage

SUMMARY:
Long-distance mountain running is increasingly popular among European and North America countries. Long-distance races are organized in various mountains and can reach up to 160 km (100 miles) with several thousands meters of climbing. The pathophysiological consequences of such extreme effort is still a matter a debate. From a muskelo-skeletal perspectives, the potential lower-limb join damage is a major health issue. The present study aims to use objective magnetic resonance imaging (MRI) techniques to describe the consequences of performing long-distance mountain running races on the knee cartilage.

DETAILED DESCRIPTION:
Healthy male runners will perform T2 MRI knee cartilage examination before, immediatly after and 1 month after 3 distinct long-distance mountain races of 40, 55 and 160 km. The physiological responses during the races (speed, heart rate, glycemia) will also be recordered.

ELIGIBILITY:
Inclusion Criteria:

* no cardiac, respiratory or neuromuscular diseases
* more than 2 years of experience in mountain race
* no contre-indication for participating in a mountain race

Exclusion Criteria:

* history of knee surgery
* contre-indication to MRI

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male runners
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
T2 MRI | from before to immediatly after the long-distance race
  Change in T2 relaxation time of the knee cartilage

SECONDARY OUTCOMES:
Heart rate | Continuous measurement during the race
  Mean heart rate during the race
Glycemia | Continuous measurement during the race
  Mean glycemia during the race

CONTACTS AND LOCATIONS:
Overall Officials: stephane Doutreleau, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Doutreleau, Grenoble, France

IPD SHARING:
Plan to Share IPD: No